CLINICAL TRIAL: NCT06984484
Title: A Multicenter, RandoMized, Double-blind, Parallel-grOup, Afluxin® Stick Pack vs. Inactive contRol Clinical Investigation to Evaluate the Performance and Safety in Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: Performance and Safety of Afluxin® in Patients With Gastroesophageal Reflux Disease
Acronym: ARMOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Devintec Sagl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DVT2024-3
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease; GERD; Afluxin
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Afluxin® (Experimental): Afluxin® is a medical device not CE marked yet. According to the Annex VIII of MDR 2017/745 it belongs to class III (Rule 21). Afluxin® stick pack is an oral suspension to be taken without any liquid 3 times a day after breakfast, lunch and before going to bed.
  Afluxin® does not contain any medicinal substances, human or animal tissues or their derivatives, or other biologically active substances coming in contact with the patient.
  The composition of one stick pack of Afluxin® is the following: purified water, isolated pea proteins, tamarind seed polysaccharide (Tamarindus indica L.), polyacrylic acid, propyl 4-hydroxybenzoate sodium salt, sodium methylparaben, strawberry aroma, mint aroma, sodium hydroxide, sucralose.
  Interventions: Device: Afluxin®
- Placebo (Placebo Comparator): Placebo is an inactive preparation designed to match the active treatment in taste and have a similar color (white-transparent) to Afluxin®.
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: Afluxin® — Afluxin® stick pack is an oral suspension to be taken without any liquid 3 times a day after breakfast, lunch and before going to bed, for 7 days.
  Arms: Afluxin®
Drug: Placebo — Inactive control stick pack is an oral suspension to be taken without any liquid 3 times a day after breakfast, lunch and before going to bed, for 7 days.
  Arms: Placebo

SUMMARY:
Gastroesophageal Reflux Disease (GERD) is a chronic condition in which stomach acid flows back into the esophagus, causing irritation and inflammation. GERD is categorized into Nonerosive Reflux Disease (NERD), Erosive Esophagitis (EE), and Barrett's esophagus (BE). Common symptoms include heartburn and acid regurgitation. Lifestyle factors such as smoking, obesity, and Helicobacter pylori infection can increase the risk of developing GERD. The clinical management of GERD typically involves Proton Pump Inhibitors (PPIs) therapy, which, although effective, may not benefit all patients and can be associated with long-term risks. The American College of Gastroenterology (ACG) suggests PPIs discontinuation or on-demand therapy for uncomplicated GERD after an 8-week trial. However, evidence indicates that PPIs are used more frequently, often long-term and in high doses, and not necessarily according to recommendations. Moreover, the availability of Over-The-Counter (OTC) PPIs has led to prolonged use by patients without medical guidance. Concerns have been raised due to potential side effects of long-term PPIs use, including enteric, respiratory, and urinary tract infections, as well as an increased risk of vitamin and mineral deficiencies and osteoporosis.

Alternatives to PPIs include Histamine-2 Receptor Antagonists (H2RAs), antacids and alginate-based formulations. Among OTC treatments, medical devices formulated with natural components are also gaining attention for their potential performance and tolerability in managing mild to moderate GERD symptoms. These alternatives could address the unmet needs of NERD patients, especially those with a low response to PPIs treatment and provide an option without the potential side effects of prolonged PPIs use. Afluxin® is a class III medical device, containing functional substances (tamarind seed polysaccharide, pea protein and polyacrylic acid), formulated for the treatment of mild to moderate GERD. Preclinical data have shown that Afluxin® is able to create a protective barrier over the gastroesophageal epithelium, preventing reflux damage. In vitro studies suggest that Afluxin® effectively binds to the esophageal and gastric mucosa, reducing abnormal permeability caused by acid reflux. Moreover, in vivo evidence shows that Afluxin® can increase gastric pH, reduce epigastric pain, esophageal damage, and inflammatory markers associated with GERD. Given the encouraging results obtained in preclinical investigations, this study is designed to provide clinical evidence to support the performance and safety of Afluxin® in reducing gastrointestinal symptoms of patients with mild to moderate GERD in a multicenter, randomized, double-blind, parallel-group, Afluxin® stick pack vs. inactive control clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, aged ≥ 18 years and ≤ 75 years.
2. Evidence of symptomatic GERD: patients with ongoing heartburn and/or regurgitation (with or without dyspepsia symptoms of epigastric pain and/or burning) of at least mild to moderate severity or experienced during the least 7 days before starting the treatment, as assessed on a clinical basis by the Investigator.
3. Patients not pre-treated with PPIs, even for problems different from GERD (e.g., gastroprotection, PPI-based triple or quadruple therapy for eradication of H. pylori), H2RAs, and/or with antiacids, alginates or medical devices made of substances (i.e., substance-based medical devices to treat GERD, gastroesophageal reflux and similar conditions) in the last week prior to screening.
4. Patient has provided written informed consent after being informed of the study procedures and risks prior to any study-related events.
5. Patients are able to understand and adhere to the study procedures.
6. Females of childbearing potential must have a negative urine pregnancy test (dipstick) at Visit 1 and currently use or agree to use consistently and correctly (i.e., perfect use) a highly effective or acceptable effective contraceptive method for the individual subject and her partner(s) throughout the study treatment period.

Exclusion Criteria:

1. Patient with hypersensitivity to any Afluxin® or inactive control components.
2. Rhinosinusitis or bronchitis.
3. Patients with a:

   1. history and/or
   2. symptom profile and/or
   3. discovered on endoscopy suggestive of the following: any other Gastrointestinal (GI) disease, erosive GERD, BE, acute peptic ulcer and/or ulcer complications, hiatus hernia with a diameter which exceeds 3 cm, Zollinger-Ellison syndrome, esophageal or gastric cancer, pyloric stenosis, esophageal or gastric surgery, intestinal obstruction, current pernicious anemia, indication for H. pylori eradication therapy, known gastro-intestinal bleeding (hematochezia or hematemesis) within the last 12 months.
4. Patients diagnosed with functional dyspepsia characterized by postprandial distress syndrome (i.e., bothersome postprandial fullness and/or early satiation).
5. Patients with a history of gastro-esophageal surgery, anti-reflux, or bariatric procedure.
6. Presence of any active malignancy (except for non-invasive basal or squamous cell carcinoma of the skin).
7. Patients using any drug that could affect symptoms or affecting the gastrointestinal tract during the last week prior to screening:

   1. prokinetics
   2. systemic glucocorticosteroids
   3. Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)
8. Patients who are pregnant or lactating.
9. Patients who are enrolled in or have participated in other clinical trials or investigations within 30 days prior to screening.
10. Clinically significant or unstable concurrent diseases whose sequelae or treatment might contraindicate study participation or interfere with the study evaluation parameters, as judged by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assess the superiority of a 7-day treatment course with Afluxin® over inactive control in terms of difference between treatment groups in terms of proportion of responders | From enrollment to the end of the 7-day treatment
  The primary endpoint is the difference between treatment groups (Afluxin® and placebo) in terms of proportion of responders, defined as patients who report a reduction in the GERD dimension of the RDQ (Reflux Disease Questionnaire) equal to 1.5 points (clinically significant difference, according to Wilkinson et al., 2019), between baseline and the end of the 7-day treatment.
  In the RDQ questionnaire validated in Italian language, patients are asked to rate GERD-related symptoms they have been experiencing over the past 7 days. The questionnaire consists of 12 items to report the frequency and severity of heartburn, regurgitation and dyspepsia. In this study the two subscales for heartburn and regurgitation will be combined into the GERD dimension. Symptom frequency and severity will be measured on 6-point scales (ranging from 0=none to 5 =daily/severe).

SECONDARY OUTCOMES:
RDQ GERD dimension, including single item scores | Baseline and at the end of the 7-day treatment
  GERD dimension evaluated through the RDQ (Reflux Disease Questionnaire) and evaluation of the single item scores, at the baseline and at the end of the 7-day treatment.
  In the RDQ questionnaire validated in Italian language, patients are asked to rate GERD-related symptoms they have been experiencing over the past 7 days. The self-assessed questionnaire will consist of 12 items to report the frequency and severity of heartburn, regurgitation and dyspepsia. The two subscales for heartburn and regurgitation will be combined into the GERD dimension. Symptom frequency and severity will be measured on 6-point scales (ranging from 0=none to 5 =daily/severe).
RDQ dyspepsia dimension total and single item scores | Baseline and at the end of the 7-day treatment
  Dyspepsia dimension evaluated through the RDQ (Reflux Disease Questionnaire) total and single item scores, at the baseline and at the end of the 7-day treatment.
  In the RDQ questionnaire validated in Italian language, patients are asked to rate GERD-related symptoms they have been experiencing over the past 7 days. The self-assessed questionnaire will consist of 12 items to report the frequency and severity of heartburn, regurgitation and dyspepsia (burning/pain in the upper stomach). Symptom frequency and severity will be measured on 6-point scales (ranging from 0=none to 5 =daily/severe).
Total and single item scores of the Reflux Symptom Index (RSI) | Baseline and at the end of the 7-day treatment
  Total and single item scores of the Reflux Symptom Index (RSI) at baseline and at the end of the 7-day treatment, assessing the severity of Laryngopharyngeal Reflux (LPR) symptoms.
  The RSI validated in Italian language, will be used for the evaluation of LPR symptoms that patients have been experiencing within the last month. The RSI examines 9 items, to be scored from 0 (no problem) to 5 (severe problem), with a higher score indicating a higher severity of the symptom (range of total score: 0-45) .
Severity of GERD cardinal symptoms (i.e., heartburn and regurgitation) | Throughout the 7-day treatment
  Severity of GERD cardinal symptoms (i.e., heartburn and regurgitation) throughout the 7-day treatment, as self-assessed daily by patients using a 7-point Likert scale ranging from 1 = no discomfort to 7 = very severe discomfort.
Severity of LPR symptoms (i.e., hoarseness/clearing the throat and troublesome cough) | Throughout the 7-day treatment
  Severity of (Laryngopharyngeal Reflux) LPR symptoms (i.e., hoarseness/clearing the throat and troublesome cough) throughout the 7-day treatment, as self-assessed daily by patients using a 7-point Likert scale ranging from 1 = no discomfort to 7 = very severe discomfort.
Number and percentage of patients with occurrence of symptoms during the night | Throughout the 7-day treatment
  Number and percentage of patients with occurrence of symptoms during the night throughout the 7-day treatment
Mean time to alleviation of symptoms following treatment administration | Throughout the 7-day treatment
  Mean time to alleviation of symptoms following treatment administration throughout the 7-day treatment, as self-assessed daily by patients
Number and percentage of patients with complete remission of symptoms | At the end of the 7-day treatment
  Number and percentage of patients with complete remission of symptoms at the end of the 7-day treatment, defined as an RDQ (Reflux Disease Questionnaire) GERD dimension total score = 0 points.
  In the RDQ questionnaire validated in Italian language, patients are asked to rate GERD-related symptoms they have been experiencing over the past 7 days. The self-assessed questionnaire will consist of 12 items to report the frequency and severity of heartburn, regurgitation and dyspepsia. Symptom frequency and severity will be measured on 6-point scales (ranging from 0=none to 5 =daily/severe).
Mean score on the self-report measure Patient's Global Impression of Change (PGI-C) | At the end of the 7-day treatment
  Mean score on the self-report measure Patient's Global Impression of Change (PGI-C) at the end of the 7-day treatment, assessing the patient's overall perceived change in their condition.
  The self-report measure PGI-C will be used to assess the overall perceived improvement at the end of the 7-day treatment. Patients will reply to the general statement "Since the start of the study, my overall status is'", using the following 7-point scale: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse.
Number and percentage of patients who take prohibited medications | Throughout the 7-day treatment
  Number and percentage of patients who take prohibited medications (Proton Pump Inhibitors, Histamine-2 Receptor Antagonists, antiacid, alginates or medical devices made of substances).
Patient's compliance with treatment | Throughout the 7-day treatment
  Patient's compliance with treatment protocol, in terms of adherence to the instructions and recommendations of the study treatment protocol. The information are recorded on the patient's diary and reviewed by the investigators. Patient differences in % compliance between the two treatments will be calculated.
Patient's satisfaction with treatment | At the end of the 7-day treatment
  Patient's satisfaction with treatment, as self-assessed by the patient using a 5-point response scale, at the end of the 7-day treatment.
  At the end of the 7-day treatment the patient will record his/her opinion of satisfaction with treatment in the e-diary, answering the question: "How satisfied are you with the study treatment you received?" with a 5-point response scale (1=unsatisfied, 2=somewhat unsatisfied, 3=neutral, 4=somewhat satisfied, 5=satisfied).
Safety: adverse events and device deficiencies | Throughout the 7-day treatment
  Incidence and type of AEs and DDs continuously monitored during the study

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - IRCCS Policlinico San Martino, Genova
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation, Milan
  - AOU Federico II di Napoli, Napoli
  - Azienda Ospedale Università Padova, Padua
  - Humanitas Research Hospital, Rozzano (MI)
  - A.O.U. Città della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: No